CLINICAL TRIAL: NCT01095757
Title: Evaluation of Plerixafor (Mozobil ™, AMD3100) in Combination With Chemotherapy and G-CSF for CD34+ Cell Mobilization
Brief Title: Evaluation of the Drug Plerixafor in Combination With Chemotherapy and G-CSF for Stem Cell Collection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Edmund Waller, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00027735; WCI1671-09 (Other: Other)
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Myeloma; Lymphoma
Keywords: Myeloma; Lymphoma; Stem cell transplantation
MeSH Terms: conditions — Neoplasms, Plasma Cell; Lymphoma | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plerixafor + Chemo and G-CSF (Other): Patients who receive a combination of Plerixafor, chemotherapy and G-CSF.
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — 240 µg/kg subcutaneous injection on the day that the absolute neutrophil count (ANC) is > 1500/mm3 and on each day of apheresis for a total of 4 aphereses or the target CD34 cell dose has been reached.
  Other Names: Mozobil; AMD3100

SUMMARY:
The purpose of this study is to test whether the addition of the drug plerixafor to treatment with chemotherapy and G-CSF can better activate your bone marrow stem cells to improve the chances of transplant. The study will look for the activation of a certain type of blood cell, called CD34+ cells in patients who receive plerixafor, chemotherapy and G-CSF. The investigators will follow the number of patients that achieve the target numbers of CD34+ cells. The number of patients achieving the target level of CD34+ cells, and the total number of CD34+ cells, will be compared to the numbers in previous studies testing just chemotherapy and G-CSF, without plerixafor.

The investigators will also test the safety of the combination of plerixafor with chemotherapy and G-CSF and look at the success of the transplantation after 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Multiple myeloma (MM) or non-Hodgkin's lymphoma (NHL) patients in first or second complete or partial remission
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Up to 3 prior treatment regimens
5. Meet all eligibility requirements for autologous transplant
6. Adequate marrow function defined as white blood cells (WBC) >3,000; ANC >1,500/mm3; platelets >75,000/mm3
7. Adequate renal function defined as creatinine clearance > 30 mL/min by Cockcroft-Gault
8. Adequate liver function defined as aspartate aminotransferase (AST)/alanine aminotransferase (ALT)/bilirubin < 2 times upper limit of normal
9. Able to provide informed consent
10. Women not pregnant and agree to use contraception

Exclusion Criteria:

1. High risk co-morbidities for acute treatment complications (e.g., symptomatic coronary artery disease)
2. Brain metastases or carcinomatous meningitis
3. Previous treatment with high dose chemotherapy and autologous transplant
4. Previous attempt to collect B-hematopoietic progenitor cells (HPCs) following mobilization with growth factors alone, growth factors and chemotherapy, or plerixafor and growth factors
5. Acute infection or unexplained fever >38°C
6. Weight > 175% of ideal body weight as defined by the Devine equation
7. Experimental therapy within 4 weeks
8. Cytokine administration in the previous 14 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Waller, MD, PhD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Background] Lazarus HM, Loberiza FR Jr, Zhang MJ, Armitage JO, Ballen KK, Bashey A, Bolwell BJ, Burns LJ, Freytes CO, Gale RP, Gibson J, Herzig RH, LeMaistre CF, Marks D, Mason J, Miller AM, Milone GA, Pavlovsky S, Reece DE, Rizzo JD, van Besien K, Vose JM, Horowitz MM. Autotransplants for Hodgkin's disease in first relapse or second remission: a report from the autologous blood and marrow transplant registry (ABMTR). Bone Marrow Transplant. 2001 Feb;27(4):387-96. doi: 10.1038/sj.bmt.1702796. PMID 11313668
- [Background] Lemoli RM, Martinelli G, Zamagni E, Motta MR, Rizzi S, Terragna C, Rondelli R, Ronconi S, Curti A, Bonifazi F, Tura S, Cavo M. Engraftment, clinical, and molecular follow-up of patients with multiple myeloma who were reinfused with highly purified CD34+ cells to support single or tandem high-dose chemotherapy. Blood. 2000 Apr 1;95(7):2234-9. PMID 10733490
- [Background] Smith TJ, Khatcheressian J, Lyman GH, Ozer H, Armitage JO, Balducci L, Bennett CL, Cantor SB, Crawford J, Cross SJ, Demetri G, Desch CE, Pizzo PA, Schiffer CA, Schwartzberg L, Somerfield MR, Somlo G, Wade JC, Wade JL, Winn RJ, Wozniak AJ, Wolff AC. 2006 update of recommendations for the use of white blood cell growth factors: an evidence-based clinical practice guideline. J Clin Oncol. 2006 Jul 1;24(19):3187-205. doi: 10.1200/JCO.2006.06.4451. Epub 2006 May 8. PMID 16682719
- [Background] Siena S, Bregni M, Brando B, Ravagnani F, Bonadonna G, Gianni AM. Circulation of CD34+ hematopoietic stem cells in the peripheral blood of high-dose cyclophosphamide-treated patients: enhancement by intravenous recombinant human granulocyte-macrophage colony-stimulating factor. Blood. 1989 Nov 1;74(6):1905-14. PMID 2478216
- [Background] Cassens U, Momkvist PH, Zuehlsdorf M, Mohr M, Kienast J, Berdel WE, Sibrowski W. Kinetics of standardized large volume leukapheresis (LVL) in patients do not show a recruitment phenomenon of peripheral blood progenitor cells (PBPC). Bone Marrow Transplant. 2001 Jul;28(1):13-20. doi: 10.1038/sj.bmt.1703082. PMID 11498739
- [Background] Koenigsmann M, Jentsch-Ullrich K, Mohren M, Becker E, Heim M, Franke A. The role of diagnosis in patients failing peripheral blood progenitor cell mobilization. Transfusion. 2004 May;44(5):777-84. doi: 10.1111/j.0041-1132.2004.03321.x. PMID 15104662
- [Background] Hicks ML, Lonial S, Langston A, Flowers C, Roback JD, Smith KJ, Mossavi Sai S, Teagarden D, Hamilton ES, Waller EK, Kaufman J. Optimizing the timing of chemotherapy for mobilizing autologous blood hematopoietic progenitor cells. Transfusion. 2007 Apr;47(4):629-35. doi: 10.1111/j.1537-2995.2007.01164.x. PMID 17381621
- [Background] Li J, Hamilton E, Vaughn L, Graiser M, Renfroe H, Lechowicz MJ, Langston A, Prichard JM, Anderson D, Gleason C, Lonial S, Flowers CR, Kaufman JL, Waller EK. Effectiveness and cost analysis of "just-in-time" salvage plerixafor administration in autologous transplant patients with poor stem cell mobilization kinetics. Transfusion. 2011 Oct;51(10):2175-82. doi: 10.1111/j.1537-2995.2011.03136.x. Epub 2011 Apr 14. PMID 21492180
- [Background] Kumar S, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Gastineau DA, Litzow MR, Fonseca R, Roy V, Rajkumar SV, Gertz MA. Impact of lenalidomide therapy on stem cell mobilization and engraftment post-peripheral blood stem cell transplantation in patients with newly diagnosed myeloma. Leukemia. 2007 Sep;21(9):2035-42. doi: 10.1038/sj.leu.2404801. Epub 2007 Jun 21. PMID 17581613
- [Background] Mazumder A, Kaufman J, Niesvizky R, Lonial S, Vesole D, Jagannath S. Effect of lenalidomide therapy on mobilization of peripheral blood stem cells in previously untreated multiple myeloma patients. Leukemia. 2008 Jun;22(6):1280-1; author reply 1281-2. doi: 10.1038/sj.leu.2405035. Epub 2007 Nov 22. No abstract available. PMID 18033320
- [Background] Paripati H, Stewart AK, Cabou S, Dueck A, Zepeda VJ, Pirooz N, Ehlenbeck C, Reeder C, Slack J, Leis JF, Boesiger J, Torloni AS, Fonseca R, Bergsagel PL. Compromised stem cell mobilization following induction therapy with lenalidomide in myeloma. Leukemia. 2008 Jun;22(6):1282-4. doi: 10.1038/sj.leu.2405100. Epub 2008 Jan 24. No abstract available. PMID 18216870
- [Background] Christopher MJ, Rao M, Liu F, Woloszynek JR, Link DC. Expression of the G-CSF receptor in monocytic cells is sufficient to mediate hematopoietic progenitor mobilization by G-CSF in mice. J Exp Med. 2011 Feb 14;208(2):251-60. doi: 10.1084/jem.20101700. Epub 2011 Jan 31. PMID 21282380
- [Background] Ponomaryov T, Peled A, Petit I, Taichman RS, Habler L, Sandbank J, Arenzana-Seisdedos F, Magerus A, Caruz A, Fujii N, Nagler A, Lahav M, Szyper-Kravitz M, Zipori D, Lapidot T. Induction of the chemokine stromal-derived factor-1 following DNA damage improves human stem cell function. J Clin Invest. 2000 Dec;106(11):1331-9. doi: 10.1172/JCI10329. PMID 11104786
- [Background] Jung Y, Wang J, Schneider A, Sun YX, Koh-Paige AJ, Osman NI, McCauley LK, Taichman RS. Regulation of SDF-1 (CXCL12) production by osteoblasts; a possible mechanism for stem cell homing. Bone. 2006 Apr;38(4):497-508. doi: 10.1016/j.bone.2005.10.003. Epub 2005 Dec 5. PMID 16337237
- [Background] DiPersio JF, Stadtmauer EA, Nademanee A, Micallef IN, Stiff PJ, Kaufman JL, Maziarz RT, Hosing C, Fruehauf S, Horwitz M, Cooper D, Bridger G, Calandra G; 3102 Investigators. Plerixafor and G-CSF versus placebo and G-CSF to mobilize hematopoietic stem cells for autologous stem cell transplantation in patients with multiple myeloma. Blood. 2009 Jun 4;113(23):5720-6. doi: 10.1182/blood-2008-08-174946. Epub 2009 Apr 10. PMID 19363221
- [Background] Kaufman JL, Flowers CR, Rados KD, Calandra GB, Vose JM, Hewes LB, Lonial S, Langston AA, Khoury HJ, Lechowicz MJ, Waller EK. A prospective clinical trial evaluating the safety and efficacy of the combination of rituximab and plerixafor as a mobilization regimen for patients with lymphoma. Transfusion. 2013 Jan;53(1):76-84. doi: 10.1111/j.1537-2995.2012.03719.x. Epub 2012 May 25. PMID 22624594

RESULTS

PARTICIPANT FLOW:
Groups:
- Plerixafor + Chemo and G-CSF: Patients who receive a combination of Plerixafor, chemotherapy and granulocyte-colony stimulating factor (G-CSF).
  Plerixafor : 240 µg/kg subcutaneous injection on the day that the absolute neutrophil count (ANC) is > 1500/mm3 and on each day of apheresis for a total of 4 aphereses or the target cluster of differentiation 34 (CD34) cell dose has been reached.
Period: Overall Study
Arm/Group | Plerixafor + Chemo and G-CSF
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Plerixafor + Chemo and G-CSF: Patients who receive a combination of Plerixafor, chemotherapy and G-CSF.
  Plerixafor : 240 µg/kg subcutaneous injection on the day that the ANC is > 1500/mm3 and on each day of apheresis for a total of 4 aphereses or the target CD34 cell dose has been reached.
Arm/Group | Plerixafor + Chemo and G-CSF
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years]
  Multiple Myeloma (MM), n = 17 | 58 [33 to 72]
  Lymphoma, n = 28 | 56 [38 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Patients Achieving Greater Than or Equal to 5 x 10^6 of CD34+ Cells/kg in a Single Day of Apheresis
Time Frame: Within the first 4 days following the first dose of Plerixafor
Measure: Number; unit: participants
Groups:
- Multiple Myeloma; Lymphoma: Patients who receive a combination of Plerixafor, chemotherapy and G-CSF.
  Plerixafor : 240 µg/kg subcutaneous injection on the day that the ANC is > 1500/mm3 and on each day of apheresis for a total of 4 aphereses or the target CD34 cell dose has been reached.
Arm/Group | Multiple Myeloma | Lymphoma
Number analyzed (Participants) | 10 | 23
participants | 9 | 17

2. Secondary Outcome: Average Number of Days for Engraftment (Engraftment Defined as Absolute Neutrophil Count>500)
Time Frame: Within the first 4 days following the first dose of Plerixafor
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Multiple Myeloma | Lymphoma
Number analyzed (Participants) | 10 | 23
days | 12.4 (1.62) | 12.105 (1.63)

3. Primary Outcome: Patients Achieving >= 3 X 10^6 CD34+ Cell/Kg
Time Frame: Within the first 4 days following the first dose of Plerixafor
Measure: Number; unit: participants
Arm/Group | Multiple Myeloma | Lymphoma
Number analyzed (Participants) | 10 | 23
participants | 10 | 23

ADVERSE EVENTS:
Arm/Group | Plerixafor + Chemo and G-CSF
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 29/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plerixafor + Chemo and G-CSF (N=45)
Nausea (Gastrointestinal disorders) | 13
Bone Pain (Musculoskeletal and connective tissue disorders) | 12
Diarrhea (Gastrointestinal disorders) | 12
Fatigue (General disorders) | 11
Hypokalemia (Blood and lymphatic system disorders) | 8
Lightheadedness (General disorders) | 7
Headache (General disorders) | 6
Thrombocytopenia Grade 1/2 (Blood and lymphatic system disorders) | 26
Thrombocytopenia Over Grade 2 (Blood and lymphatic system disorders) | 17
Anemia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes